CLINICAL TRIAL: NCT03922750
Title: A Trial Comparing NNC0148-0287 C (Insulin 287) Versus Insulin Glargine U100, Both in Combination With Metformin, With or Without DPP4 Inhibitors and With or Without SGLT2 Inhibitors, in Basal Insulin Treated Subjects With Type 2 Diabetes Mellitus
Brief Title: A Research Study in People With Type 2 Diabetes to Compare Two Types of Insulin: Insulin 287 and Insulin Glargine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN1436-4466; U1111-1219-5541 (Other: World Health Organization (WHO)); 2018-003407-18 (EudraCT Number)
Record Dates: First submitted 2019-04-17; First posted 2019-04-22 (Actual); Results first posted 2021-01-08 (Actual); Last update posted 2022-01-18 (Actual); Status verified 2022-01

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — insulin icodec

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Insulin 287 (with 100% loading dose) (Experimental): Participants will receive insulin 287 injections once weekly (OW). A unit to unit switch approach with an additional 100% loading dose of insulin 287 will be used.
  Interventions: Drug: Insulin icodec
- Insulin 287 (without loading dose) (Experimental): Participants will receive insulin 287 injections OW. A unit to unit switch approach without loading dose of insulin 287 will be used.
  Interventions: Drug: Insulin icodec
- Insulin glargine U100 (Active Comparator): Participants will receive insulin glargine U100 once daily (OD).
  Interventions: Drug: Insulin glargine U100

INTERVENTIONS:
Drug: Insulin icodec — Participants will receive subcutaneous (s.c.) injections of Insulin 287 OW for 16 weeks.
  Other Names: Insulin 287
  Arms: Insulin 287 (with 100% loading dose); Insulin 287 (without loading dose)
Drug: Insulin glargine U100 — Participants will receive s.c. injections of insulin glargine OD for 16 weeks
  Arms: Insulin glargine U100

SUMMARY:
This study compares insulin 287 (a possible new medicine) to insulin glargine (a medicine doctors can already prescribe) in people with type 2 diabetes. Different ways of switching from the insulin which the participants are already on to insulin 287 are also compared. This is done to find the best way to switch to insulin 287. The participants will either get insulin 287 that they will have to inject once a week or insulin glargine that they will have to inject once a day. Which treatment any participant gets is decided by chance. The study will last for about 5 months (23 weeks). The participants will have 14 clinic visits and 6 phone calls with the study doctor. At 3 of the clinic visits participants will be asked not to eat or drink anything (except for water) in the last 8 hours before the visit. During the study, the doctor will ask the participants to: 1) measure their blood sugar every day with a blood sugar meter using a finger prick; 2) write down different information in a diary daily and return this to their study doctor. 3) wear a medical device (sensor) that measures the participants blood sugar all the time for 18 weeks (about 4 months) during the study.

ELIGIBILITY:
Inclusion criteria:

* Male or female, aged 18-75 years (both inclusive) at the time of signing informed consent.
* Diagnosed with type 2 diabetes mellitus greater than or equal to 180 days prior to the day of screening.
* Glycosylated haemoglobin (HbA1c) of 7.0-10.0% (53.0-85.8 mmol/mol) (both inclusive) as assessed by central laboratory.
* Treated with once daily or twice daily basal insulin analogue (insulin degludec, insulin detemir, insulin glargine U100 or U300, total daily dose of 10-50 U, both inclusive) greater than or equal to 90 days prior to the day of screening.
* Stable daily dose(s) for 90 days prior to the day of screening of any of the following antidiabetic drug(s) or combination regime(s):

  1. Any metformin formulations greater than or equal to 1500 mg or maximum tolerated or effective dose (as documented in subject's medical records).
  2. Free or fixed combination therapy: Metformin as outlined above with or without dipeptidyl peptidase 4 inhibitors (DPP4i) with or without sodium-glucose cotransporter 2 inhibitors (SGLT2i) is allowed: 1) DPP4i (greater than or equal to half of the maximum approved dose according to local label or maximum tolerated or effective dose); 2) SGLT2i (greater than or equal to half of the maximum approved dose according to local label or maximum tolerated or effective dose.
* Body mass index (BMI) less than or equal to 40.0 kg/m^2.

Exclusion criteria:

* Known or suspected hypersensitivity to trial product(s) or related products.
* Female who is pregnant, breast-feeding or intends to become pregnant or is of child-bearing potential and not using an adequate contraceptive method.
* Participation in any clinical trial of an approved or non-approved investigational medicinal product within 90 days before screening.
* Any disorder, except for conditions associated with type 2 diabetes mellitus, which in the investigator's opinion might jeopardise subject's safety or compliance with the protocol.
* Any episodes of diabetic ketoacidosis within the past 90 days prior to the day of screening and between screening and randomisation.
* Known hypoglycaemic unawareness as indicated by the Investigator according to Clarke's questionnaire question 8.
* Recurrent severe hypoglycaemic episodes within the last year as judged by the Investigator.
* Myocardial infarction, stroke, hospitalisation for unstable angina pectoris or transient ischaemic attack within 180 days prior to the day of screening and between screening and randomisation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2019-05-09 (Actual); Primary Completion 2019-12-19 (Actual); Study Completion 2020-01-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Reporting Anchor and Disclosure (1452), Study Director — Novo Nordisk A/S
Locations (33):
- United States (9):
  - Novo Nordisk Investigational Site, Walnut Creek, California
  - Novo Nordisk Investigational Site, Roswell, Georgia
  - Novo Nordisk Investigational Site, Idaho Falls, Idaho
  - Novo Nordisk Investigational Site, Las Vegas, Nevada
  - Novo Nordisk Investigational Site, Nashua, New Hampshire
  - Novo Nordisk Investigational Site, Chattanooga, Tennessee
  - Novo Nordisk Investigational Site, Nashville, Tennessee
  - Novo Nordisk Investigational Site, Dallas, Texas
  - Novo Nordisk Investigational Site, Renton, Washington
- Canada (10):
  - Novo Nordisk Investigational Site, Edmonton, Alberta
  - Novo Nordisk Investigational Site, Surrey, British Columbia
  - Novo Nordisk Investigational Site, Vancouver, British Columbia
  - Novo Nordisk Investigational Site, Halifax, Nova Scotia
  - Novo Nordisk Investigational Site, Brampton, Ontario
  - Novo Nordisk Investigational Site, Concord, Ontario
  - Novo Nordisk Investigational Site, Etobicoke, Ontario
  - Novo Nordisk Investigational Site, Hamilton, Ontario
  - Novo Nordisk Investigational Site, Markham, Ontario
  - Novo Nordisk Investigational Site, Sarnia, Ontario
- Czechia (4):
  - Novo Nordisk Investigational Site, Broumov
  - Novo Nordisk Investigational Site, Holešov
  - Novo Nordisk Investigational Site, Hranice
  - Novo Nordisk Investigational Site, Trutnov
- Germany (6):
  - Novo Nordisk Investigational Site, Falkensee
  - Novo Nordisk Investigational Site, Hamburg
  - Novo Nordisk Investigational Site, Ludwigshafen
  - Novo Nordisk Investigational Site, Münster
  - Novo Nordisk Investigational Site, Oldenburg I. Holst
  - Novo Nordisk Investigational Site, Saint Ingbert-Oberwürzbach
- Italy (4):
  - Novo Nordisk Investigational Site, Bergamo
  - Novo Nordisk Investigational Site, Catanzaro
  - Novo Nordisk Investigational Site, Milan
  - Novo Nordisk Investigational Site, Roma

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com

REFERENCES:
- [Result] Bajaj HS, Bergenstal RM, Christoffersen A, Davies MJ, Gowda A, Isendahl J, Lingvay I, Senior PA, Silver RJ, Trevisan R, Rosenstock J. Switching to Once-Weekly Insulin Icodec Versus Once-Daily Insulin Glargine U100 in Type 2 Diabetes Inadequately Controlled on Daily Basal Insulin: A Phase 2 Randomized Controlled Trial. Diabetes Care. 2021 Jul;44(7):1586-1594. doi: 10.2337/dc20-2877. Epub 2021 Apr 19. PMID 33875485

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 34 sites in 5 countries as follows: Canada (10), Italy (5), Czech Republic (4), Germany (5) and the United States (10). In addition, 3 sites in the United states and 1 site in Germany screened, but didn't randomise any subjects.
Pre-assignment Details: Participants were randomised to receive once weekly insulin 287 using any of 2 different switch approaches or once daily insulin glargine; as an add-on to background therapy with basal insulin analogue with metformin, with or without dipeptidyl peptidase-4 inhibitors (DPP4i) and with or without sodium-glucose cotransporter 2 inhibitors (SGLT2i) at stable, pre-trial dose and at same frequency during the entire treatment period unless due to safety concerns related to the background medication.
Groups:
- Insulin 287 (Without Loading Dose): Participants were to receive once weekly subcutaneous (s.c.) injection of insulin 287 for 16 weeks, using PDS290 prefilled pen-injector at a starting dose of 7 times the pre-trial basal insulin dose of the respective participants ('unit to unit switch' approach: current daily dose x 7). Participants were to perform once daily pre-breakfast self-monitoring plasma glucose (SMPG). The dose was adjusted based on 3 pre-breakfast SMPG values measured on the 2 previous days and the day of the contact. If at least one pre-breakfast SMPG value was: < 4.4 millimoles per litre (mmol/L): dose reduced by 28 U; 4.4-7.2 mmol/L: no adjustment; > 7.2 mmol/L: dose increased by 28 U. If the participant received a twice-daily regimen with any basal insulin analogue or a once-daily regimen with insulin glargine U300 prior to randomisation, the total daily insulin dose prior to randomisation was reduced by 20%.
- Insulin 287 (With 100% Loading Dose): Participants were to receive once weekly s.c. injection of insulin 287 for 16 weeks, using PDS290 prefilled pen-injector at a starting dose of 7 times the pre-trial basal insulin dose of the respective participants with additional loading dose ('unit to unit switch with an additional 100% loading dose' approach: current daily dose x 7 x 2). Participants were to perform once daily pre-breakfast SMPG. The dose was adjusted based on 3 pre-breakfast SMPG values measured on the 2 previous days and the day of the contact. If at least one pre-breakfast SMPG value was: < 4.4 millimoles per litre (mmol/L): dose reduced by 28 U; 4.4-7.2 mmol/L: no adjustment; > 7.2 mmol/L: insulin dose increased by 28 U. If the participant received a twice-daily regimen with any basal insulin analogue or a once-daily regimen with insulin glargine U300 prior to randomisation, the total daily insulin dose prior to randomisation was reduced by 20%.
- Insulin Glargine U100: Participants were to receive once daily s.c. injection of insulin glargine U100 for 16 weeks, using SoloSTAR prefilled pen-injector at a starting dose same as the pre-trial basal insulin. Participants were to perform once daily pre-breakfast SMPG. The dose was adjusted based on 3 pre-breakfast SMPG values measured on the 2 previous days and the day of the contact. If at least one pre-breakfast SMPG value was: < 4.4 millimoles per litre (mmol/L): dose reduced by 4 U; 4.4-7.2 mmol/L: no adjustment; > 7.2 mmol/L: insulin dose increased by 4 U. If the participant received a twice-daily regimen with any basal insulin analogue or a once-daily regimen with insulin glargine U300 prior to randomisation, the total daily insulin dose prior to randomisation was reduced by 20%.
Period: Overall Study
Arm/Group | Insulin 287 (Without Loading Dose) | Insulin 287 (With 100% Loading Dose) | Insulin Glargine U100
Started | 50 | 54 | 50
Full Analysis Set (FAS) | 50 | 54 | 50
Safety Analysis Set (SAS) | 50 | 54 | 50
Completed | 50 | 53 | 49
Not Completed | 0 | 1 | 1
Not completed — Unclassified | 0 | 0 | 1
Not completed — Adverse Event | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The full analysis set included all randomised participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Insulin 287 (Without Loading Dose) | Insulin 287 (With 100% Loading Dose) | Insulin Glargine U100 | Total
Number analyzed (Participants) | 50 | 54 | 50 | 154
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.1 (8.2) | 62.4 (7.2) | 60.5 (7.9) | 61.7 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 15 | 17 | 43
  Male | 39 | 39 | 33 | 111
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 6 | 6 | 13
  Not Hispanic or Latino | 49 | 48 | 44 | 141
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 9 | 4 | 3 | 16
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Black or African American | 2 | 3 | 3 | 8
  White | 39 | 46 | 44 | 129
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Time in Target Range 3.9-10.0 mmol/L (70-180 Milligrams Per Deciliter (mg/dL)) Measured Using CGM (Continuous Glucose Monitoring)
Description: The percentage of time spent in glycaemic target range was calculated as 100 times the number of recorded measurements in glycaemic target range 3.9-10.0 mmol/L (70-180 mg/dL), both inclusive divided by the total number of recorded measurements. The endpoint was evaluated based on the data from the on-treatment without rescue medication observation period, which was the time period when a participant was on treatment with trial product, excluding any period after initiation of a non-randomised insulin treatment (rescue medication).
Time Frame: During the last 2 weeks of treatment (week 15 and 16)
Population: Full analysis set included all randomised participants. Overall number of participants analyzed = participants with available data.
Measure: Least Squares Mean (Standard Error); unit: Percentage of time
Arm/Group | Insulin 287 (Without Loading Dose) | Insulin 287 (With 100% Loading Dose) | Insulin Glargine U100
Number analyzed (Participants) | 49 | 53 | 50
Percentage of time | 65.99 (2.34) | 72.86 (2.13) | 64.98 (2.23)
Statistical Analysis 1: Comparison: Insulin 287 (Without Loading Dose) vs Insulin Glargine U100; The response and change from baseline in response during last two weeks of treatment (week 15 and 16) were analysed using an analysis of covariance (ANCOVA) model with treatment, pre-trial insulin treatment and SGLT2i use as fixed factors, and baseline response as covariate. Missing endpoint values were imputed using multiple imputation based on own treatment arm with baseline response as a covariate. Each imputed dataset was analysed separately and estimates were combined using Rubin's rules; Test type: Other; p = 0.7542, ANCOVA; Estimated mean treatment difference = 1.01, 95% CI 2-sided [-5.33 to 7.35]
Statistical Analysis 2: Comparison: Insulin 287 (With 100% Loading Dose) vs Insulin Glargine U100; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.0107, ANCOVA; Estimated mean treatment difference = 7.88, 95% CI 2-sided [1.83 to 13.93]

2. Secondary Outcome: Change in Glycosylated Haemoglobin (HbA1c)
Description: Estimated mean change from baseline (week 0) in HbA1c at week 16 is presented. The endpoint was evaluated based on the data from the on-treatment without rescue medication observation period, which was the time period when a participant was on treatment with trial product, excluding any period after initiation of a non-randomised insulin treatment (rescue medication).
Time Frame: From baseline week 0 (V2) to week 16 (V18)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percentage point of HbA1c
Arm/Group | Insulin 287 (Without Loading Dose) | Insulin 287 (With 100% Loading Dose) | Insulin Glargine U100
Number analyzed (Participants) | 50 | 54 | 50
Percentage point of HbA1c | -0.47 (0.09) | -0.77 (0.09) | -0.54 (0.09)

3. Secondary Outcome: Change in Fasting Plasma Glucose (FPG)
Description: Estimated mean change from baseline (week 0) in FPG at week 16 is presented. The endpoint was evaluated based on the data from the on-treatment without rescue medication observation period, which was the time period when a participant was on treatment with trial product, excluding any period after initiation of a non-randomised insulin treatment (rescue medication).
Time Frame: From baseline week 0 (V2) to week 16 (V18)
Population: Full analysis set included all randomised participants. Overall number analyzed = participants with available data.
Measure: Least Squares Mean (Standard Error); unit: Millimoles per liter (mmol/L)
Arm/Group | Insulin 287 (Without Loading Dose) | Insulin 287 (With 100% Loading Dose) | Insulin Glargine U100
Number analyzed (Participants) | 50 | 52 | 49
Millimoles per liter (mmol/L) | -0.83 (0.23) | -0.69 (0.22) | -0.57 (0.23)

4. Secondary Outcome: Change in Body Weight
Description: Estimated mean change from baseline (week 0) in body weight at week 16 is presented. The endpoint was evaluated based on the data from the on-treatment without rescue medication observation period, which was the time period when a participant was on treatment with trial product, excluding any period after initiation of a non-randomised insulin treatment (rescue medication).
Time Frame: From baseline week 0 (V2) to week 16 (V18)
Population: Full analysis set included all randomised participants. Overall number analyzed = participants with available data.
Measure: Least Squares Mean (Standard Error); unit: Kilogram (Kg)
Arm/Group | Insulin 287 (Without Loading Dose) | Insulin 287 (With 100% Loading Dose) | Insulin Glargine U100
Number analyzed (Participants) | 50 | 54 | 50
Kilogram (Kg) | 1.32 (0.36) | 0.61 (0.34) | 0.10 (0.35)

5. Secondary Outcome: Weekly Insulin Dose
Description: Estimated mean average weekly insulin dose during the last 2 weeks of treatment is presented. The endpoint was evaluated based on the data from the on-treatment without rescue medication observation period, which was the time period when a participant was on treatment with trial product, excluding any period after initiation of a non-randomised insulin treatment (rescue medication).
Time Frame: During the last 2 weeks of treatment (week 15 and 16)
Population: Full analysis set included all randomised participants. Overall Number analyzed = participants with available data.
Measure: Least Squares Mean (95% Confidence Interval); unit: Units of insulin (U)
Arm/Group | Insulin 287 (Without Loading Dose) | Insulin 287 (With 100% Loading Dose) | Insulin Glargine U100
Number analyzed (Participants) | 50 | 54 | 50
Units of insulin (U) | 242.31 [205.49 to 285.74] | 191.03 [163.06 to 223.81] | 195.91 [166.19 to 230.94]

6. Secondary Outcome: Number of Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event(AE) is any untoward medical occurrence in a clinical trial subject administered or using a medicinal product, whether or not considered related to the medicinal product or usage.. A TEAE was defined as an event that had onset date (or increase in severity) during the on-treatment observation period. The on-treatment observation period was the time period from first dose of trial product until the follow-up visit or the last date on trial product + 5 weeks for once daily insulin and +6 weeks for once weekly insulin. Safety analysis set (SAS) included all subjects exposed to at least one dose of trial product.
Time Frame: From baseline week 0 (V2) to week 21 (V20)
Population: Safety analysis set (SAS) included all participants exposed to at least one dose of trial product.
Measure: Number; unit: Count of events
Arm/Group | Insulin 287 (Without Loading Dose) | Insulin 287 (With 100% Loading Dose) | Insulin Glargine U100
Number analyzed (Participants) | 50 | 54 | 50
Count of events | 77 | 85 | 76

7. Secondary Outcome: Number of Severe Hypoglycaemic Episodes (Level 3)
Description: Severe hypoglycaemic episodes (level 3) were defined as episodes that were associated with severe cognitive impairment requiring external assistance for recovery. Number of severe hypoglycaemic episodes that occurred during weeks 0-16 are presented.
Time Frame: From baseline week 0 (V2) to week 16 (V18)
Population: SAS included all participants exposed to at least one dose of trial product.
Measure: Number; unit: Count of events
Arm/Group | Insulin 287 (Without Loading Dose) | Insulin 287 (With 100% Loading Dose) | Insulin Glargine U100
Number analyzed (Participants) | 50 | 54 | 50
Count of events | 0 | 0 | 0

8. Secondary Outcome: Number of Clinically Significant Hypoglycaemic Episodes (Level 2) (Below 3.0 mmol/L (54 mg/dL), Confirmed by BG Meter) or Severe Hypoglycaemic Episodes (Level 3)
Description: Clinically significant hypoglycaemic episodes (level 2) were defined as episodes that were sufficiently low to indicate serious, clinically important hypoglycaemia with plasma glucose value of <3.0 mmol/L (54 mg/dL). Severe hypoglycaemic episodes (level 3) were defined as episodes that were associated with severe cognitive impairment requiring external assistance for recovery. Number of clinically significant hypoglycaemic episodes (level 2), confirmed by blood glucose (BG)meter or severe hypoglycaemic episodes (level 3) that occured during weeks 0-16 are presented.
Time Frame: From baseline week 0 (V2) to week 16 (V18)
Population: SAS included all participants exposed to at least one dose of trial product.
Measure: Number; unit: Count of events
Arm/Group | Insulin 287 (Without Loading Dose) | Insulin 287 (With 100% Loading Dose) | Insulin Glargine U100
Number analyzed (Participants) | 50 | 54 | 50
Count of events | 3 | 17 | 16

9. Secondary Outcome: Number of Hypoglycaemic Alert Episodes(Level 1) (Greater Than or Equal to 3.0 and Below 3.9 mmol/L (Greater Than or Equal to 54 and Below 70 mg/dL), Confirmed by BG Meter)
Description: Hypoglycaemia alert value (level 1) was defined as episodes that were sufficiently low for treatment with fast-acting carbohydrate and dose adjustment of glucose-lowering therapy. Number of hypoglycaemic alert episodes (level 1) (equal to or above 3.0 and below 3.9 mmol/L (equal to or above 54 and below 70 mg/dL), confirmed by BG meter) that occured during weeks 0-16 are presented.
Time Frame: From baseline week 0 (V2) to week 16 (V18)
Population: SAS included all participants exposed to at least one dose of trial product.
Measure: Number; unit: Count of events
Arm/Group | Insulin 287 (Without Loading Dose) | Insulin 287 (With 100% Loading Dose) | Insulin Glargine U100
Number analyzed (Participants) | 50 | 54 | 50
Count of events | 79 | 78 | 71

ADVERSE EVENTS:
Time Frame: Weeks 0-21.
Description: Results are based on the safety analysis set which included all participants exposed to at least one dose of trial product. All presented adverse events are TEAEs. TEAE was defined as an event that had onset date (or increase in severity) during the on-treatment observation period.
Arm/Group | Insulin 287 (Without Loading Dose) | Insulin 287 (With 100% Loading Dose) | Insulin Glargine U100
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/54 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50 | 2/54 | 1/50
Other Adverse Events (participants affected / at risk) | 18/50 | 20/54 | 18/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin 287 (Without Loading Dose) (N=50) | Insulin 287 (With 100% Loading Dose) (N=54) | Insulin Glargine U100 (N=50)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Muscle abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin 287 (Without Loading Dose) (N=50) | Insulin 287 (With 100% Loading Dose) (N=54) | Insulin Glargine U100 (N=50)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 4 (4)
Diabetic retinopathy (Eye disorders) | 2 (2) | 2 (2) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 3 (4)
Headache (Nervous system disorders) | 1 (1) | 3 (3) | 3 (3)
Hypertension (Vascular disorders) | 3 (3) | 1 (1) | 1 (1)
Influenza (Infections and infestations) | 3 (3) | 1 (1) | 0 (0)
Instillation site haemorrhage (General disorders) | 0 (0) | 0 (0) | 4 (7)
Medical device site haemorrhage (General disorders) | 2 (2) | 5 (7) | 1 (3)
Nasopharyngitis (Infections and infestations) | 7 (8) | 8 (9) | 2 (3)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (4) | 1 (1) | 1 (2)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property.

DOCUMENTS (2):
  • Study Protocol (2020-05-28): https://cdn.clinicaltrials.gov/large-docs/50/NCT03922750/Prot_000.pdf
  • Statistical Analysis Plan (2020-05-28): https://cdn.clinicaltrials.gov/large-docs/50/NCT03922750/SAP_001.pdf